CLINICAL TRIAL: NCT00615615
Title: Evaluation of the Efficacy and Tolerability of Levetiracetam Add-On Treatment in Refractory Pediatric Patients With Partial Onset Seizures: A 28-Week Double-Blind, Placebo-Controlled Multi-center Trial
Brief Title: Efficacy and Tolerability of Levetiracetam Add-On Treatment in Refractory Pediatric Patients With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: UCB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N159
Record Dates: First submitted 2008-01-27; First posted 2008-02-14 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (LEV) (Experimental): LEV dose was titrated to a level of 60 mg/kg/day. The initial dose level was 20 mg/kg/day for the first two weeks, followed by a dose level of 40 mg/kg/day for two weeks. If lower doses were well tolerated, the LEV dose was increased to a dose level of 60 mg/kg/day for the remaining 10 weeks. The dose level could be reduced to 40 mg/kg/day if the patient did not tolerate LEV at a dose level of 60 mg/kg/day.
  Interventions: Drug: Levetiracetam
- Placebo (Placebo Comparator): Subjects received Placebo matching to LEV treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — * high total tablet weight (HTTW) formulation in tablet strengths of 166.5 mg, 250 mg, and 500 mg was used for patients weighing at least 40.1 kg
  * low total tablet weight (LTTW) formulation in tablet strengths of 166 mg and 250 mg was used for patients weighing 40 kg or less
  Arms: Levetiracetam (LEV)
Drug: Placebo — Placebo tablets for oral administration that were identical in appearance to the respective formulations (LTTW and HTTW) were used as reference therapy
  Arms: Placebo

SUMMARY:
Double-blind, randomized, placebo-controlled, multi-center clinical trial conducted to evaluate levetiracetam as adjunctive therapy in children (4-16 years) with refractory partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of epilepsy with uncontrolled partial onset seizures, whether or not secondarily generalized, and the diagnosis was >= 6 months before the Selection Visit
* epilepsy was classifiable according to the ILAE Classification
* >= 4 partial onset seizures during the 4 weeks preceding the Selection Visit and were required to have >= 4 partial onset seizures during each 4-week interval of the Baseline Period to qualify for randomization
* unsatisfactory current AED treatment in terms of efficacy and/or safety
* stable AED treatment consisting of no more than two AEDs

Exclusion Criteria:

* treatable seizure etiology
* epilepsy secondary to a progressive cerebral disease or any other progressively neurodegenerative disease, including Rasmussen and Landau-Kleffner diseases
* history of status epilepticus which required hospitalization during 3 months prior to the Selection Visit
* history of or the presence of pseudo seizures
* current diagnosis of Lennox-Gastaut syndrome

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 1999-09 (Actual); Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Partial onset seizure frequency (Type I, Type IC included) per week during the Treatment period | During the 14-weeks Treatment period (Week 8 to Week 22)
  Calculated as 7-day partial onset seizure frequency.

SECONDARY OUTCOMES:
50% responder rate in seizure frequency per week during the Treatment Period | During the 14-weeks Treatment period (Week 8 to Week 22)
  Response rate is defined as percent of patients experiencing at least a 50% reduction from baseline in the seizure frequency per week during the Treatment Period.
Percent of patients with categorized reduction from baseline in seizure frequency per week during the Treatment Period | From Baseline to the 14-weeks Treatment period
  Categories as follows: <-25%, -25% to <25%, 25% to <50%, 50% to <75%, 75% to <100%, and 100%
Change from baseline in the average duration of seizure free intervals | From Baseline to the 14-weeks Treatment period
  Intervals are defined as seizure-free if no seizures are reported.
Number of seizure free days during the Treatment Period | During the 14-weeks Treatment period (Week 8 to Week 22)
  A day is regarded as seizure-free if no seizures are reported.
Absolute change from baseline in partial onset seizure frequency per week during the Treatment Period | Baseline, During the 14-weeks Treatment period (Week 8 to Week 22)
  Absolute change from baseline in partial onset seizure frequency during the Treatment Period standardized to 1 week period.
  A negative value in absolute change from baseline indicates a decrease in partial onset seizure frequency from baseline.
Absolute change from baseline in partial onset seizure frequency per week during the Titration Period | Baseline, During the 6-weeks Titration period (Week 8 to Week 14)
  Absolute change from baseline in partial onset seizure frequency during the Titration Period standardized to 1 week period.
  A negative value in absolute change from baseline indicates a decrease in partial onset seizure frequency from baseline.
Absolute change from baseline in partial onset seizure frequency per week during the Evaluation Period | Baseline, During the 8-weeks Evaluation period (Week 14 to Week 22)
  Absolute change from baseline in partial onset seizure frequency during the Evaluation Period standardized to 1 week period.
  A negative value in absolute change from baseline indicates a decrease in partial onset seizure frequency from baseline.
Percent change from baseline in partial onset seizure frequency per week during the Treatment Period | Baseline, During the 14-weeks Treatment period (Week 8 to Week 22)
  Percent change from baseline in partial onset seizure frequency during the Treatment Period standardized to 1 week period.
  A negative value in absolute change from baseline indicates a decrease in partial onset seizure frequency from baseline.
Percent change from baseline in partial onset seizure frequency per week during the Titration Period | Baseline, During the 6-weeks Titration period (Week 8 to Week 14)
  Percent change from baseline in partial onset seizure frequency during the Titration Period standardized to 1 week period.
  A negative value in absolute change from baseline indicates a decrease in partial onset seizure frequency from baseline.
Percent change from baseline in partial onset seizure frequency per week during the Evaluation Period | Baseline, During the 8-weeks Evaluation period (Week 14 to Week 22)
  Percent change from baseline in partial onset seizure frequency during the Evaluation Period standardized to 1 week period.
  A negative value in absolute change from baseline indicates a decrease in partial onset seizure frequency from baseline.
Cumulative percentage of patients who were seizure-free since the beginning of the Evaluation Period | Beginning of the Evaluation Period (Week 14)
  A subject was regarded as seizure-free if not seizures were reported since the beginning of the Evaluation Period.
Partial onset seizure frequency per week during the Titration Period | During the 6-weeks Titration period (Week 8 to Week 14)
  Calculated as 7-day partial onset seizure frequency.
Partial onset seizure frequency per week during the Evaluation Period | During the 6-weeks Evaluation period (Week 8 to Week 14)
  Calculated as 7-day partial onset seizure frequency.
Total seizure frequency per week (Types I + II + III) during the Treatment Period | During the 14-weeks Treatment period (Week 8 to Week 22)
  Calculated as 7-day partial onset seizure frequency.
Total seizure frequency per week (Types I + II + III) during the Titration Period | During the 6-weeks Titration period (Week 8 to Week 14)
  Calculated as 7-day partial onset seizure frequency.
Total seizure frequency per week (Types I + II + III) during the Evaluation Period | During the 6-weeks Evaluation period (Week 8 to Week 14)
  Calculated as 7-day partial onset seizure frequency.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)

REFERENCES:
- [Background] Glauser TA, Ayala R, Elterman RD, Mitchell WG, Van Orman CB, Gauer LJ, Lu Z; N159 Study Group. Double-blind placebo-controlled trial of adjunctive levetiracetam in pediatric partial seizures. Neurology. 2006 Jun 13;66(11):1654-60. doi: 10.1212/01.wnl.0000217916.00225.3a. Epub 2006 Apr 26. PMID 16641323
- [Background] Jensen FE, Bourgeois BF. Randomized trial supports use of levetiracetam adjunctive therapy to treat partial seizures in children. Nat Clin Pract Neurol. 2006 Nov;2(11):596-7. doi: 10.1038/ncpneuro0325. No abstract available. PMID 17057745
- [Derived] Johnson ME, McClung C, Bozorg AM. Analyses of seizure responses supportive of a novel trial design to assess efficacy of antiepileptic drugs in infants and young children with epilepsy: Post hoc analyses of pediatric levetiracetam and lacosamide trials. Epilepsia Open. 2021 Jun;6(2):359-368. doi: 10.1002/epi4.12482. Epub 2021 May 3. PMID 34033237